CLINICAL TRIAL: NCT02154152
Title: A CLINICAL STUDY TO EVALUATE THE EFFICACY OF CAUSTICUM 200C IN THE TREATMENT OF PRIMARY ENURESIS
Brief Title: A Clinical Study on Causticum 200 Centesimal Potency in Primary Enuresis
Acronym: PE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fr Muller Homoeopathic Medical College (Other)
Collaborators: Father Muller Medical College (Other)
Responsible Party: Principal Investigator, Jyoshna Shivaprasad, Dr Jyoshna Shivaprasad, Fr Muller Homoeopathic Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: enuresishmc
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Bed Wetting; Primary Enuresis
Keywords: Bed wetting; Primary Enuresis; Frequency; Efficacy; Homoeopathic Medicine; Causticum 200c
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Homoeopathic Medicine Causticum (Experimental): The drug namely Causticum 200C potency shall be administered as 4 globules, prescribed once a week for 3 months with placebo to follow for the remaining period.
  Interventions: Drug: Homoeopathic Medicine causticum 200c

INTERVENTIONS:
Drug: Homoeopathic Medicine causticum 200c
  Other Names: Potassium Hydrate, Hahnemann's Tinctura Acris Sine Kali

SUMMARY:
Homeopathic Medicine Causticum 200c will be prescribed in cases of Primary Enuresis on the basis of available symptoms for a period of one year and the results will be evaluated at the end of the given period and efficacy of the drug will be assessed.

DETAILED DESCRIPTION:
A CLINICAL STUDY TO EVALUATE THE EFFICACY OF CAUSTICUM 200C IN THE TREATMENT OF PRIMARY ENURESIS

AIMS & OBJECTIVES:

To assess and evaluate the efficacy of administering the Homoeopathic remedy Causticum 200 Centesimal potency based on Homoeopathic principles in management of Primary enuresis A total number of 30 cases will be selected after screening 50 cases as per the inclusion criteria from the Outpatient Department of Father Muller Homoeopathic Medical College for the study and will be followed for a period of one year.

Inclusion criteria:

1. Age group between 5-15 yrs
2. Both sexes are included
3. Patients with Primary enuresis will be Included
4. Patients with Nocturnal or Diurnal enuresis will be included

Exclusion criteria:

1 Patients with metabolic illness like Diabetes Mellitus or Diabetes Insipidus will be excluded 2. Congenital anomalies like horse shoe kidney, polycystic kidney will be excluded.

3. Presence of Malignancy, Mental Retardation and Cerebral palsy will be excluded.

The case shall be analyzed and prescribed the remedy Causticum in 200 Centesimal potency, 4 globules once a week for 3 months with placebo to follow for the next few months and general management.

RESEARCH PLAN:

Purposive sampling will be followed in the study wherein patients who belong to the above category of Inclusion criteria will be taken up and subjected to screening so as to confirm the diagnosis of Enuresis.

Each patient will be treated for one year with Causticum 200C in the first 3 months along with placebo to follow and attended to, once a week. At each follow-up they will be assessed clinically for evaluating the improvement status.

The drug namely Causticum 200C potency will be ordered from Father Muller Homoeopathic Pharmaceutical division, which complies with the standards of Homoeopathic Pharmacopeia of India. The dosage shall be 4 globules prescribed once a week for 3 months with placebo to follow for the remaining period. This medicine shall be advised half an hour before food.

RESEARCH METHODOLOGY AND STATISTICS:

Criteria for deciding the Efficacy of Homoeopathic medicine Causticum200C shall be based on the following parameters:

1. Frequency of Enuresis
2. Odor of urine
3. Diurnal and Nocturnal urination
4. Modalities

PLAN FOR ANALYSIS: The collected data will be analyzed by paired 't' test to determine the efficiency.

RESEARCH HYPOTHESIS: There is significant improvement among Primary Enuresis cases in Paediatric age group after prescribing the Homoeopathic drug Causticum 200C.

NULL HYPOTHESIS: There is no significant improvement among Primary Enuresis cases in Paediatric age group after prescribing the Homoeopathic drug Causticum 200C.

ALTERNATIVE HYPOTHESIS: Significant variation in the above parameters before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* • Age group between 5-15 yrs

  * Both sexes are included
  * Patients with Primary enuresis will be Included
  * Patients with Nocturnal or Diurnal enuresis will be included

Exclusion Criteria:

* •Patients with metabolic illness like Diabetes Mellitus or Diabetes Insipidus will be excluded

  * Congenital anomalies like horse shoe kidney, polycystic kidney will be excluded.
  * Presence of Malignancy, Mental Retardation and Cerebral palsy will be excluded.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Bring down frequency of bed wetting | 1month
  The patients with nocturnal enuresis will receive causticum 200c on weekly basis and results expected by one month.

CONTACTS AND LOCATIONS:
Overall Officials: Jyoshna Shivaprasad, MD (Hom), Principal Investigator — Father Muller Homoeopathic Medical College
Locations (1):
- Father Muller Homoeopathic Medical College, Mangalore, Karnataka, India